CLINICAL TRIAL: NCT00766974
Title: Compression Versus Anti-Embolism Stockings in Patients With Leg Edema: Objective Investigation of Interface Compression and Edema Measurements, Clinical Outcomes, and Quality of Life.
Brief Title: Compression Aided Management of Edema in Patients With C3 Venous Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BSN Medical Inc (Industry)
Responsible Party: Joseph D. Raffetto, MD, Boston VA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSNCL-0003
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Venous Disease
Keywords: Chronic Venous Disease; C3; Edema; Compression Garments; Compression Stockings; Bioimpedance
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Anti-embolism Knee High compression stocking
  Interventions: Device: Anti-embolism Knee High Stocking
- 2 (Active Comparator): 20-30mmHg Knee High Jobst Compression Stocking
  Interventions: Device: 20-30 Knee High Compression Stocking

INTERVENTIONS:
Device: Anti-embolism Knee High Stocking — Anti-embolism Knee High Compression Stocking
  Other Names: Kendall TEDS
  Arms: 1
Device: 20-30 Knee High Compression Stocking — 20-30 mmHg Knee High COmpression Stocking
  Other Names: Jobst 20-30 mmHg Compression Stocking
  Arms: 2

SUMMARY:
Objectives: To quantify the clinical improvement and quality of life between patients wearing compression stockings versus anti-embolism stockings in patients with varicose veins and limb edema.

DETAILED DESCRIPTION:
Research Design: Pilot study of patients presenting to vascular clinic with chronic venous disease with varicose veins and/or edema will be randomized 1:1 in one of two compression garment groups. Measurements of edema and the interface compression applied at the ankle will be determined. The venous clinical severity scoring system and quality of life are assessed. After 4 weeks of treatment patients will have repeat objective studies and clinical outcomes determined.

Methodology: Patients with venous disease and edema and non-venous edema will be evaluated by clinical exam and venous duplex ultrasound. Patients eligible for the study will be randomized to knee-high 20-30 Hg graded compression stockings or anti-embolism (13-18 mm Hg) compression stockings. Patients will have limb quantitative edema assessment, a severity score and quality of life determination. Compression will be assigned to each treatment group with instruction on proper wear and duration, and the interface pressure of compression at the skin surface at the ankle level determined. Following 4 weeks of compression, patients will return for evaluation in the following areas: quantify limb edema, quantify compression at the ankle, venous clinical severity score, and venous disease specific quality of life. Data will be analyzed and presented as mean±sd. Data are analyzed using ANOVA followed by Scheffe's F test for comparison of multiple means. Student's t-test for unpaired and paired data will be used for comparison of two means. Differences are considered statistically significant if P < 0.05.

Significance: Utilizing objective measures of leg edema and applied interface pressure with two different compression garments, the data will provide the important relation between compression (mm Hg) and function of an appropriate graded compression stocking in improving limb edema and symptoms. In addition, measuring clinical outcomes before and after compression will validate the usefulness of proper compression. This study is intended to identify important quantifiable parameters that may be useful in assessing treatment end point including: clinical improvement, length of treatment, daily treatment utilization, prognosis, and clinical guidelines for compression in a specific clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with varicose veins exhibiting lower leg edema
* Unilateral or bi-lateral edema

Exclusion Criteria:

* Generalized leg edema from renal disease, heart failure, liver disease or other undetermined cause
* Acute infection
* Hepatitis
* Steroid use
* immuno-deficiencies including HIV
* Acute deep venous thrombosis
* Have had leg surgery or other orthopedic procedure in past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Edema reduction measured by bio-impedance | 4 weeks

SECONDARY OUTCOMES:
Clinical Venous Severity Score Improvement in QOL | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Raffetto, MD, Principal Investigator — Boston VA Healthcare
Locations (1):
- Boston VA Healthcare, West Roxbury, Massachusetts, United States